CLINICAL TRIAL: NCT03758521
Title: Natural History Study of Patients With Succinic Semialdehyde Dehydrogenase (SSADH) Deficiency
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Washington State University (Other); University of South Florida (Other); University Hospital Heidelberg (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Phillip Pearl, Director of Epilepsy and Clinical Neurophysiology, William G. Lennox Chair, Boston Children's Hospital, Boston Children's Hospital
Other Study IDs: IRB-P00029917; 1R01HD091142-01A1 (NIH)
Record Dates: First submitted 2018-11-16; First posted 2018-11-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Succinic Semialdehyde Dehydrogenase Deficiency
Keywords: SSADHD; SSADH deficiency
MeSH Terms: conditions — succinic semialdehyde dehydrogenase deficiency | interventions — Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio-specimen collection will include blood, urine, saliva, hair, stool, and a skin biopsy. Blood, urine, saliva, blood spots, and hair samples will also be banked for to-be-determined (TBD) studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BCH Cohort: Patients enrolled at BCH will travel to BCH every 2 years at a minimum for comprehensive evaluation taking place over a 48 hour period. Visits to BCH may occur within ± 2 months of the scheduled visit date. Electronic surveys will be sent out every 6 months.Visits will consist of clinical assessments (demographics, medical history, physical examination, neurological exam, medication history, neuropsychological assessments, and clinical severity score), neurophysiological assessments (Brain Magnetic resonance imaging [MRI/MRS/DTI], Electroencephalogram [EEG], and Transcranial magnetic stimulation [TMS]), and yearly bio-specimen collection.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Device: Magnetic resonance imaging (MRI); Device: Electroencephalogram (EEG); Procedure: Bio-specimen Collection
- iNTD Cohort: Patients enrolled at iNTD sites will travel to their iNTD site according to standard of care requirements. Data collection includes clinical history and relevant laboratory-chemical, therapeutic, instrumental and neuropsychological parameters by the study centers. Data collection takes place within the framework of elective outpatient visits. The collected parameters are congruent with the current standard investigations. Electronic surveys will be sent out every 6 months. Imaging and neurophysiological data will be collected if performed during the clinical visit or if performed as part of the site's ongoing research. Yearly bio-specimen collection will be attempted after consent is obtained from the family.
  Interventions: Procedure: Bio-specimen Collection
- Standard of Care Cohort: Patients enrolled at other sites will attend their visit at their regular clinical site as mandated by standard of care. Data collection includes medical history, family history, medications, and all clinical and neuropsychological assessments listed. Imaging and neurophysiological data will be collected if performed during the clinical visit or if performed as part of the clinical site's ongoing research. Yearly bio-specimen collection will be attempted.
  Interventions: Procedure: Bio-specimen Collection

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a method for noninvasive electrical cortical stimulation, where small intracranial currents are generated by a powerful, fluctuating, extracranial magnetic field. TMS is unique in its capacity for experimental, diagnostic, and therapeutic utility. Single pulse (spTMS) and paired-pulse TMS (ppTMS) have been used extensively to study, measure, and modulate cortical excitability and plasticity.
  Other Names: Nexstim Navigated Brain Stimulation (NBS) System 4
  Groups: BCH Cohort
Device: Magnetic resonance imaging (MRI) — These will be outpatient MRI studies that are planned without sedation. Subjects enrolled at BCH will undergo brain MRI, including volumetric MRI, MRS, and diffusion tensor imaging (DTI). The data will help define the natural history of brain volume, brain myelination and spectroscopic (e.g. GABA) abnormalities.
  Groups: BCH Cohort
Device: Electroencephalogram (EEG) — These will be outpatient EEG recordings that span 20-60 minutes and done without sedation. Recordings will be performed using electrode locations specified by the international 10-20 system for standard clinical practice.
  Other Names: Natus
  Groups: BCH Cohort
Procedure: Bio-specimen Collection — Bio-specimen collection will include blood, urine, saliva, hair, stool, and a skin biopsy. Blood, urine, saliva, blood spots, and hair samples will also be banked for to-be-determined (TBD) studies.

SUMMARY:
Succinic Semialdehyde Dehydrogenase deficiency (SSADHD) is a rare autosomal recessive disease that interferes with the catabolism of the major inhibitory neurotransmitter gamma-amino butyric acid (GABA) and furthermore leads to accumulation of various potential toxic metabolites, most prominently gamma hydroxybutyric acid (GHB). Current research indicates that there is developmental delay and significant neurophysiological and biochemical alterations in SSADHD patients, but whether disease presentation varies with age is not known. The investigators propose to determine the natural course of the clinical presentation of SSADHD; to determine the natural course of neurophysiological and biochemical indices known to be altered in SSADHD; and to identify neurophysiological and biochemical predictors of clinical severity.

The overall objective is to define the natural course of the clinical, neurophysiological and biochemical spectrum of SSADHD. Secondary objectives include the identification of biomarkers that correlate with disease phenotype and predict clinical outcomes, and the creation of an international SSADHD data repository for future investigation of pathogenesis and therapy.

DETAILED DESCRIPTION:
The study will be conducted by 4 academic institutions: Washington State University (WSU), Boston Children's Hospital (BCH), University of South Florida (USF), and University Children's Hospital Heidelberg (iNTD). The design of the study is mixed, with longitudinal and cross-sectional assessments over a period of 5 years.

Patients will be separated into three cohorts. The Boston Children's cohort will be a total of 20 patients evaluated at Boston Children's Hospital in the United States. These patients will be followed for five years, and attend a visit to the hospital in years 1,3 and 5 where assessments including history/physical, neuropsychological testing, EEG, TMS, and bio-specimen collection will be completed. Each patient will have an MRI of the brain done with special GABA sequencing one time over the five years. Each visit will take place over the course of two days. At BCH, the goal will be to schedule visits every other year with questionnaires and surveys sent out up to every 6 months, and bio-specimen collection every year. The BCH team will also ask for two follow up phone calls occurring 12 months after each onsite visit. Visits will consist of clinical assessments (demographics, medical history, physical examination, neurological exam, medication history, neuropsychological assessments, and clinical severity score), neurophysiological assessments (Brain MRI/MRS/DTI, Electroencephalogram, and Transcranial magnetic stimulation), and yearly bio-specimen collection (blood, urine, saliva, hair, stool, and skin biopsy). Bio-specimens will be sent to Washington State University for testing and addition to a biorepository. The iNTD (international NeuroTransmitters Disorders) cohort will be comprised of 15 patients who are seen at European sites who will have approval through their ethics committee to share de-identified information. Bio-specimens will be attempted to be collected at each visit from patients and sent to Washington State University. At the iNTD sites and for patients followed outside of iNTD, visits and bio-specimen collections will depend on the patients' follow-up schedules with electronic, web-based survey sent on a regular schedule (every 6 months). The standard of care cohort will be comprised of 10 patients throughout the world who provide consent to share de-identified information to the database.

The data will be stored in a database on the University of South Florida server. The server is password protected, and each member of the study personal will have a unique log in to have access to the site. Subjects will also be given specialized access to complete follow up electronic web based surveys twice a year over the course of 5 years. The team at USF will assist with data analysis.

ELIGIBILITY:
Inclusion Criteria:

* 4-hydroxybutyric aciduria (γ-hydroxybutyric aciduria)
* documented pathogenic ALDH5A1 (aldehyde dehydrogenase 5A1 gene) mutation
* 0-99 years

Exclusion Criteria:

* active or recent substance abuse or dependence within the past year.
* inability to participate in the study procedures.
* any condition that makes the study subject, in the opinion of the investigator, unsuitable for the study.
* patients will be excluded from the MRI section of the study if they have: implanted cardiac pacemaker or autodefibrillators, implanted neural pacemakers, cochlear implants, metallic foreign bodies in the eye or Central Nervous System (CNS), any implanted wire or metal device that may concentrate radio frequency fields.
* patients less than age two years will be excluded from the TMS procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults diagnosed with Succinic Semialdehyde Dehydrogenase (SSADH) deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Severity Score | 5 Years
  A composite score ranging from 5 (profound impairment) to 25 (no impairment) will be calculated using scores from five clinically significant subdomains (cognition, communication, motor skills, psychiatric presentation, and epilepsy), each scored from 1 (worse) to 5 (no impairment).
Biochemical - GABA measurement | 5 Years
  GABA is measured by electron-capture negative-ion mass fragmentography. The level will be measured in the different bio-specimens.
Biochemical - GHB measurement | 5 Years
  GHB is measured using gas chromatography-mass spectrometry (GCMS). GHB will be measured in the different bio-specimens.
Quantification of GABA related signals on the MRI spectroscopy | 5 Years
  MRI spectroscopy with special editing for GABA-related peaks in multi-voxel MRS. Concentrations will be analyzed.

OTHER OUTCOMES:
Quantification of EEG abnormalities (%) | 5 Years
  Degree of epileptiform abnormalities will be recorded using the American Clinical Neurophysiology Society guidelines [Continuous (>90%), Abundant (50-89%), Frequent (10-49%), Occasional (1-9%), and Rare (< 1 %)].
Extent of altered signal hyperintensities on structural MRI (%) | 5 years
  Altered T2 and FLAIR signal hyperintensities will be reported as a percent.
Degree of myelination on structural MRI (%) | 5 years
  Degree of myelination will be reported as a percent.
Total cerebral volume on structural MRI (cm3) | 5 years
  Total cerebral volume will be reported in cubic centimeters (cm3).
Amplitudes of motor evoked potentials (mm) | 5 years
  Intracortical Inhibition (ICI) and Facilitation (ICF) are a paired-pulse TMS measure of cortical excitability. A short Interval interstimuli (2ms) leads to a cortical inhibition, which reflects the GABAergic neurotransmission; whereas a longer interval interstimuli leads to a cortical facilitation, which reflects glutamatergic neurotransmission. Analyzed by obtaining peak-to-peak amplitudes in millimeters (mm).
Durations of cortical silent period (ms) | 5 years
  Cortical Silent Period (CSP) is a single-pulse TMS measure of cortical inhibition, stimulations are applied while subjects are exerting a muscular contraction and lead to a muscular cancellation. Duration of this silence is measured in milliseconds (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Phillip L Pearl, MD, Study Chair — Boston Children's Hospital/Harvard Medical School; K. Michael Gibson, PhD, Study Chair — Washington State University
Locations (4):
- Boston Children's Hospital, Boston, Massachusetts, United States
- University Children's Hospital, Heidelberg, Heidelberg, Germany
- Sant Joan de Deu Hospital Barcelona, Barcelona, Spain
- Birmingham Children's Hospital NHS Foundation Trust, Birmingham, United Kingdom

REFERENCES:
- [Derived] Tokatly Latzer I, Lee HHC, Yang E, Alves C, Bertoldi M, Fung C, Steele SV, Kule E, Jin Z, Rotenberg A, Roullet JB, Pearl PL. Central Dysmyelination in SSADH-Deficient Humans and Mice. Ann Clin Transl Neurol. 2025 Nov;12(11):2193-2205. doi: 10.1002/acn3.70148. Epub 2025 Jul 31. PMID 40741980
- [Derived] Tokatly Latzer I, Roullet JB, Afshar-Saber W, Lee HHC, Bertoldi M, McGinty GE, DiBacco ML, Arning E, Tsuboyama M, Rotenberg A, Opladen T, Jeltsch K, Garcia-Cazorla A, Julia-Palacios N, Gibson KM, Sahin M, Pearl PL. Clinical and molecular outcomes from the 5-Year natural history study of SSADH Deficiency, a model metabolic neurodevelopmental disorder. J Neurodev Disord. 2024 Apr 24;16(1):21. doi: 10.1186/s11689-024-09538-9. PMID 38658850